CLINICAL TRIAL: NCT04653740
Title: Omic Technologies to Track Resistance to Palbociclib in Metastatic Breast Cancer (OMERIC): A Cohort Study
Brief Title: Omic Technologies to Track Resistance to Palbociclib in Metastatic Breast Cancer
Acronym: OMERIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Laboratoire PRISM - Michel SALZET (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OMERIC-1904
Record Dates: First submitted 2020-09-15; First posted 2020-12-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Advanced Breast Cancer
Keywords: breast cancer; omics profiles; proteomics; volatile organic compounds; exosomes
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: specimen sample collection — Before and during treatment, and at progression, collection of :
  * Blood
  * Exhaled air
  * Saliva
  * Sweat
  * Tears
  * Urine

SUMMARY:
This is a monocentric cohort study, prospective and interventional with minimal risks and constraints for advanced breast cancer. The planned interventions are collection of biological samples at different times. The study will aim to do a descriptive analysis of omics profiles evolution (tumor, volatile organic components) over time, before and after disease progression under Palbociclib treatment with a clinical-biological database.

DETAILED DESCRIPTION:
Patients enrolled in the study will receive the following interventions:

* Biospecimen sample collection: before and during treatment, and at progression
* Tumor biopsy before treatment and at progression

The aim of this study is to describe molecular changes associated with resistance to Palbociclib at the individual level and describe longitudinal changes in the profile of tumor, VOCs and exosomes according to treatment response.

Other objectives of the study include:

* Proportion of single or shared molecular alterations / signatures between patients at progression time
* Associations between tumor signatures, VOCs and exosomes
* Compare molecular changes identified by proteomics with those observed by genomics / transcriptomics
* Compare the evolution of VOCs and exosomes over time with evolution of liquid biopsy markers.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* With histologically proven breast cancer, positives hormones receptors and negative HER2
* Advanced disease (metastases or non-resequable locoregional disease), from the 1st to the 4th line.
* With an indication for hormone therapy associated with the CDK4/6 inhibitor Palbociclib
* Agree to the sampling of the study
* Signed the informed consent form

Exclusion Criteria:

* Neoadjuvant or adjuvant treatment for localized breast cancer
* Metastatic breast cancer beyond the forth line
* Impossibility to give informed consent (person deprived of liberty or under guardianship)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with breast cancer
Enrollment: 25 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Intrapatient variation in molecular profiles at progression compared to baseline | From date of inclusion until the date of first documented progression (around 2 years)
  Variation over time in the rate of VOCs in response to treatment and in progression situations.
longitudinal changes in VOCs profile and exosomes according to response to treatment | From date of inclusion until the date of first documented progression, assessed up to 2 years
  variation over time in exosomes count in response to treatment and in progression situations

SECONDARY OUTCOMES:
Proportion of alterations / molecular signatures unique or shared between patients at progression | At progression time, up to 2 years
  Frequency of molecular alterations in the population
Correlation between tumor signatures, VOCs and exosomes | At progression time, up to 2 years
  Distribution of VOCs and exosome profiles according to the different molecular profiles of tumors that will be identified

OTHER OUTCOMES:
Concordance between molecular changes identified by proteomics and those observed by genomics/transcriptomics | At progression time, up to 2 years
  Concordance between identified proteins and expressed genes and/or detected mutations
Describe the evolution of VOCs and exosomes over time in relation to the evolution of liquid biopsy markers (CA15.3) | At progression time, up to 2 years
  Intra-patient variation over time in VOC rate (rate of CA15.3)
Describe the evolution of VOCs and exosomes over time in relation to the evolution of liquid biopsy markers (CA15.3) | At progression time, up to 2 years
  Intra-patient variation over time in exosomes count (rate of CA15.3)
Describe the evolution of VOCs and exosomes over time in relation to the evolution of liquid biopsy markers (CA15.3) | At progression time, up to 2 years
  Intra-patient variation over time in liquid biopsy markers (rate of CA15.3)
Describe the evolution of VOCs and exosomes over time in relation to the evolution of liquid biopsy markers (LDH) | At progression time, up to 2 years
  Intra-patient variation over time in VOC rate (rate of LDH)
Describe the evolution of VOCs and exosomes over time in relation to the evolution of liquid biopsy markers (LDH) | At progression time, up to 2 years
  Intra-patient variation over time in exosomes count (rate of LDH)
Describe the evolution of VOCs and exosomes over time in relation to the evolution of liquid biopsy markers (LDH) | At progression time, up to 2 years
  Intra-patient variation over time in liquid biopsy markers (rate of LDH)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: Yes